CLINICAL TRIAL: NCT00577265
Title: An Observational Study to Investigate How Patients Experience the Ability to Adjust Their Asthma Maintenance Medication According to Instructions Received From Their Physician (AMD).
Brief Title: An Observational Study to Investigate How Patients Experience the Ability to Adjust Their Asthma Maintenance Medication
Acronym: INVOLVE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: S43
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma Control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational study to investigate how patients experience the ability to adjust their asthma maintenance medication according to instructions received from their physician. The primary aim is to create an insight in the perception of the patient when he has the ability to adjust his own maintenance treatment and how the patient exercises this in the daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: patients with prescription of budesonide/formoterol Turbuhaler 200/6 (adjustable maintenance dosing) and whom received instructions from their physician to adjust their asthma maintenance medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Dates: Start 2004-11

PRIMARY OUTCOMES:
The primary aim is to create an insight in the perception of the patient when he has the ability to adjust his own maintenance treatment and how the patient exercises this in the daily practice.

SECONDARY OUTCOMES:
The secondary goal is to investigate the efficacy of the treatment with budesonide/formoterol AMD on the patients asthma control measured with the ACQ.

CONTACTS AND LOCATIONS:
Overall Officials: Hannie de Munnik, Study Director — AstraZeneca; Monique Scholtes, Study Chair — AstraZeneca